CLINICAL TRIAL: NCT01338701
Title: A Randomized Exploratory Study to Evaluate Two Acupuncture Methods for the Treatment of Headaches Associated With Traumatic Brain Injury
Brief Title: Exploratory Study to Evaluate 2 Acupuncture Methods for the Treatment of Headaches Associated With TBI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Samueli Institute for Information Biology (Other)
Collaborators: Defense Centers of Excellence for Psychological Health and Traumatic Brain Injury (U.S. Federal Agency); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 350890
Record Dates: First submitted 2011-03-28; First posted 2011-04-19 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Headache; Traumatic Brain Injury
Keywords: TBI; Headaches; Military; Acupuncture; Walter Reed Army Medical Center; Fort Belvoir Community Hospital
MeSH Terms: conditions — Headache; Brain Injuries, Traumatic | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Auricular (Ear) Acupuncture (Experimental): Auricular (Ear) Acupuncture is administered in a step-wise, algorithmic acupuncture approach in which needles are inserted at specific auricular landmarks. The sequence and location of needled points is determined by the participant's severity of headache pain at presentation and response to needling. Between six and nine points are needled in each treatment session depending on the individual's response (i.e., a decrease or persistence of headache pain). In-dwelling ASP needles are inserted at the end of each session. Participants are instructed to remove the needles after 3 days, or sooner if pain or redness developed at a needle site. Ten 45-minute acupuncture treatment sessions are administered over 6 weeks.
  Interventions: Procedure: Auricular (Ear) Acupuncture
- Traditional Chinese Acupuncture (TCA) (Experimental): A semi-standardized form of Traditional Chinese Acupuncture (TCA) is administered, incorporating the insertion of up to 22 acupuncture needles associated with each individual participant's: (1) primary headache pattern (up to three pairs of points); (2) secondary headache pattern (up to 2 pairs of points); (3) Ah-Shi or tender points (up to 4 points); (4) constitutional points (source points on two meridians); and, (5) up to 2 pairs of additional points from a selected list. Point selection was reassessed every two weeks per TCM diagnostic and treatment principles. While the majority of points were located on the limbs, points also included local points of tenderness to the head, as well as the front and back of the torso. Ten 60-minute TCA sessions are administered over 6 weeks.
  Interventions: Procedure: Traditional Chinese Acupuncture (TCA)
- Usual Care (Other): All study participants continue to receive routine usual care for their TBI, headaches and associated symptoms as determined by their clinical team.
  Interventions: Other: Usual Care

INTERVENTIONS:
Procedure: Traditional Chinese Acupuncture (TCA) — An acupuncturist will examine and evaluate subjects before inserting thin, sterile stainless steel needles at specific points on their body. Patients will receive 10 treatments over a 6 week period.
  Arms: Traditional Chinese Acupuncture (TCA)
Procedure: Auricular (Ear) Acupuncture — An acupuncturist will insert sterile stainless steel needles and an ASP ear needle into various points in subject's outer ear. The ASP is a shorter needle that will stay in the participant's ear for a few days. Patients will receive 10 treatments over a 6 week period.
  Arms: Auricular (Ear) Acupuncture
Other: Usual Care — Subjects do not receive acupuncture during the 6 week study time period. Instead, they continue to receive medical care for headaches and other symptoms. They can elect to receive up to 10 ear acupuncture treatments between the 6- and 12-week assessments.
  Arms: Usual Care

SUMMARY:
This study investigates whether acupuncture can help to decrease the number and severity of headaches in people who have Traumatic Brain Injury. The aim of this study is to compare two different types of acupuncture-either Traditional Chinese Acupuncture or ear acupuncture-to a group that receives no acupuncture at all. Acupuncture has been demonstrated to reduce pain, improve health-related quality of life, prevent migraine headaches, and improve tension and chronic daily headaches.

DETAILED DESCRIPTION:
This is a 12 week study. If eligible, participants will be randomly assigned to 1of 3 groups: ear acupuncture, Traditional Chinese Acupuncture, or the usual care group.

Subjects receiving acupuncture will:

* meet with one of the acupuncturists who will conduct her first assessment
* come to Walter Reed Army Medical Center (WRAMC) 10 times over a 6-week period to receive acupuncture treatments from a licensed acupuncturist

Subjects in the usual care group will:

* not receive any acupuncture treatments
* continue usual treatment plan
* be given the option to receive 10 acupuncture treatments between the 6- and 12-week period

All subjects will also:

* complete questionnaires at 3 different times: baseline (beginning of study), after 6 weeks, and after 12 weeks. These questionnaires will assess headaches, overall health and quality of life
* complete a daily headache diary
* continue to be treated for their headaches
* continue taking prescription and over-the-counter medications for any conditions being treated

ELIGIBILITY:
Inclusion Criteria:

1. 18-69 years of age
2. Service Members with previous deployment to war zone
3. Non-acute mild to moderate traumatic brain injury as defined by:

   * Injury event (i.e., blast, fall, MVC, head impact) that occurred at least 7 days prior
   * Loss of consciousness (if present) for less than 24 hours and alteration of consciousness or posttraumatic amnesia for less than one week
4. Presence of headache or any etiology requiring self-medication or medical management with at least 4 headache days in the past 4 weeks
5. Rancho Los Amigos Cognitive Scale score of greater than or equal to 7
6. Able to provide informed consent

Exclusion Criteria:

1. Acupuncture treatment for any reason within the past month
2. Any active unstable psychiatric condition, including active psychosis, suicidal or homicidal ideation
3. Unwillingness on the part of the participant to complete all study visits and/or components of the intervention
4. Scheduled surgery during the treatment phase of the study
5. Pregnancy or breastfeeding at time of study enrollment or during study participation
6. Any medically unstable condition that in the opinion of the P.I. has the potential to warrant inpatient treatment in the medical or intensive care units
7. Inability to give informed consent or complete study measures

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Headache Impact Test at Week 6 | Baseline, Week 6, Week 12
  This is a 6-item measure that assesses headache severity. This will take approximately 1 minute to complete.

SECONDARY OUTCOMES:
Daily Headache Diary | Completed daily for 6 weeks
  Before bedtime, participants will note whether or not they had a headache that day. If they experienced a headache, they will rate it's severity and whether or not they took any medications for the headache. It takes less than a minute to complete.
Change from Baseline in Numerical Rating Scale at Week 6 | Baseline, Week 6
  This assesess pain along a 0-10 scale. It takes less than a minute to complete.
Change from Baseline in Beck Depression Inventory at Week 6 | Baseline, Week 6
  This is a 21-question inventory that rates depressive symptoms. It takes approximately 5 minutes to complete.
Change from Baseline in State-Trait Anxiety Inventory at Week 6 | Baseline, Week 6
  This is a 40-item survey that measures anxiety symptoms. It takes approximately 5 minutes to complete.
Change from Baseline in Post-Traumatic Stress Checklist (Civilian Version) at Week 6 | Baseline, Week 6
  Participants will indicate the degree to which they have experienced PTSD symptoms on a 5-point scale during the past month. It takes approximately 5 minutes to complete.
Change from Baseline in Symptom Checklist 90-R at Week 6 | Baseline, Week 6
  This is a 90-item checklist that evaluates a broad range of symptoms and psychological symptoms. It takes approximately 15 minutes to complete.
Change from Baseline in Medical Outcome Study Quality of Life at Week 6 | Baseline, Week 6
  This measure evaluates physical and psychological functioning. It takes approximately 10 minutes to complete.
Change from Baseline in Automated Neuropsychological Assessment Metrics at Week 6 | Baseline, Week 6
  This measure evaluates cognitive function and takes approximately 30 minutes to complete.
Change from Baseline in Pittsburgh Sleep Quality of Life at Week 6 | Baseline, Week 6
  This measure evaluates sleep quality and disturbances over athe past month. It takes approximately 7 minutes to complete.
Change from Baseline in Expectancy Scale at Week 6 | Baseline, Week 6
  This measures participants' pre-conceived expectations about the effect of acupuncture on headaches. It takes less than a minute to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Louis M French, PsyD, Principal Investigator — Walter Reed Army Medical Center; Heechin Chae, MD, Principal Investigator — Fort Belvoir Community Hospital
Locations (2):
- United States (2):
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Fort Belvoir Community Hospital, Alexandria, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Results will be shared in a published manuscript.